CLINICAL TRIAL: NCT06094738
Title: A Phase 1, Randomized, Open-Label, Single-Dose, Three-Way Crossover Study to Evaluate The Effect of Food on the Oral Bioavailability of Relacorilant in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Food on the Oral Bioavailability of Relacorilant in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CORT125134-129
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Relacorilant under fasted conditions (Experimental): Subjects will receive oral relacorilant 400 mg (4 X 100 mg softgel capsules) single dose on Day 1 under fasted conditions. The study period in which a subject will receive this treatment will be determined by random assignment to 1 of 6 treatment sequences.
  Interventions: Drug: Relacorilant under fasted conditions
- Relacorilant after a high-fat meal (Experimental): Subjects will receive oral relacorilant 400 mg (4 X 100 mg softgel capsules) single dose on Day 1 after a high-fat meal. The study period in which a subject will receive this treatment will be determined by random assignment to 1 of 6 treatment sequences.
  Interventions: Drug: Relacorilant after a high-fat meal
- Relacorilant after a low-fat meal (Experimental): Subjects will receive oral relacorilant 400 mg (4 X 100 mg softgel capsules) single dose on Day 1 after a low-fat meal. The study period in which a subject will receive this treatment will be determined by random assignment to 1 of 6 treatment sequences.
  Interventions: Drug: Relacorilant after a low-fat meal

INTERVENTIONS:
Drug: Relacorilant under fasted conditions — Oral relacorilant 400 mg (4 X 100 mg softgel capsules) single dose on Day 1 under fasted conditions
  Other Names: CORT125134
  Arms: Relacorilant under fasted conditions
Drug: Relacorilant after a high-fat meal — Oral relacorilant 400 mg (4 X 100 mg softgel capsules) single dose on Day 1 after a high-fat meal
  Other Names: CORT125134
  Arms: Relacorilant after a high-fat meal
Drug: Relacorilant after a low-fat meal — Oral relacorilant 400 mg (4 X 100 mg softgel capsules) single dose on Day 1 after a low-fat meal
  Other Names: CORT125134
  Arms: Relacorilant after a low-fat meal

SUMMARY:
The primary objective of the study is to evaluate the effects of a high-fat meal and of a low-fat meal on the bioavailability of relacorilant in healthy subjects.

DETAILED DESCRIPTION:
Enrolled healthy male and female subjects will be randomized to receive 1 of 6 treatment sequences, each consisting of 3 treatments in 3 periods, in a crossover design. The 3 treatments will be a single oral dose of relacorilant 400 mg 1) under fasted conditions, 2) after a high-fat meal, and 3) after a low-fat meal. Each period will last 5 days, and a 7-day washout will follow Periods 1 and 2. Blood samples will be collected predose and at serial timepoints up to 4 days (Day 5) after dosing in each period for evaluation of the bioavailability of relacorilant. Secondary objectives of the study will be evaluation of the bioavailability of relacorilant metabolites, and evaluation of safety and tolerability of relacorilant when administered to healthy subjects under fasted and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >18.5 and <30.0 kg/m^2 and body weight ≥50.0 kg for male subjects and ≥45.0 kg for female subjects
* Healthy, as defined by the absence of clinically significant illness and/or surgery within 4 weeks prior to dosing, and the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease
* Female subjects of childbearing potential who are sexually active with a non-sterile male partner must be willing to use an acceptable contraceptive method as defined in the protocol, throughout the study.
* Male subjects who are not vasectomized for at least 6 months, and who are sexually active with a female partner of childbearing potential must be willing to use an acceptable contraceptive method as defined in the protocol, from the first study drug administration until at least 90 days after the last study drug administration
* Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
* Capable of, and have given, written informed consent
* Willing to consume a high-fat breakfast, including pork
* Able to and willing to fast for any laboratory evaluations.

Exclusion Criteria:

* Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for HIV, hepatitis B, or hepatitis C
* Female subject with a positive pregnancy test at Screening
* Male subject with a pregnant partner at Screening
* Positive urine drug screen or urine cotinine test or alcohol breath test at Screening
* History of allergic reactions to relacorilant or other related drugs, or to any excipient in the formulation
* Clinically significant electrocardiogram abnormalities or vital sign abnormalities at Screening
* History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 83 mL of wine 12%, 200 mL of beer 5%, or 25 mL of alcohol 40%])
* History of significant drug abuse within 1 year prior to Screening or use of soft drugs within 3 months prior to Screening or hard drugs within 1 year of Screening
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration
* Use of medications for the timeframes specified in the protocol, with the exception of acceptable hormonal contraceptives and medications exempted by the Investigator, with agreement by the Sponsor because they are judged unlikely to affect the pharmacokinetic profile of the study drug or subject safety
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing
* Have a condition that may be aggravated by glucocorticoid antagonism (eg, asthma, any chronic inflammatory condition). Subjects with inactive seasonal hay fever may be included. Subjects with childhood (aged less than 18 years) asthma may be included provided they have had no symptoms and required no treatment for at least 5 years.
* History of malabsorption syndrome or previous gastrointestinal surgery, which could affect drug absorption or metabolism, with the exception of appendectomy and cholecystectomy
* Pregnant or breast-feeding
* Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to the last observed concentration of plasma relacorilant (AUC0-t) | Predose and at serial timepoints up to 4 days (Day 5) after dosing on Day 1
Area under the concentration-time curve from time zero extrapolated to infinity of plasma relacorilant (AUC0-inf) | Predose and at serial timepoints up to 4 days (Day 5) after dosing on Day 1
Maximal observed concentration of plasma relacorilant (Cmax) | Predose and at serial timepoints up to 4 days (Day 5) after dosing on Day 1

SECONDARY OUTCOMES:
AUC0-t of relacorilant plasma metabolites | Predose and at serial timepoints up to 4 days (Day 5) after dosing on Day 1
AUC0-inf of relacorilant plasma metabolites | Predose and at serial timepoints up to 4 days (Day 5) after dosing on Day 1
Cmax of relacorilant plasma metabolites | Predose and at serial timepoints up to 4 days (Day 5) after dosing on Day 1
Number of subjects with one or more adverse events | Up to Day 28
Number of subjects with one or more serious adverse events | Up to Day 55
Number of subjects with one or more adverse events leading to study drug discontinuation | Up to Day 25

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Custodio, Study Director — Corcept Therapeutics
Locations (1):
- inVentiv Health Clinical Research Services LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No